CLINICAL TRIAL: NCT01338428
Title: Sexual Assault Resistance Education for University Women: A Trial in Three Canadian Universities
Brief Title: Sexual Assault Resistance Education for University Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Windsor (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Charlene Y. Senn, Professor, University of Windsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MOP-110976
Record Dates: First submitted 2011-04-13; First posted 2011-04-19 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Sexual Assault
Keywords: rape; sexual assault; intervention; female university students

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brochure (Active Comparator)
  Interventions: Behavioral: Brochure
- Enhanced AAA Sexual Assault Education (Experimental)
  Interventions: Behavioral: Enhanced AAA Sexual Assault Resistance Education

INTERVENTIONS:
Behavioral: Enhanced AAA Sexual Assault Resistance Education — Resistance Program: 4x3-hour units. Unit 1 (Assess) accurate assessment of sexual assault risk. Provides: empirically-based information on situational and (male) behavioural danger cues; practice identifying risk and counteracting it. Unit 2 'Acknowledge[ment]' of risk when present. Includes: women's sexual rights; emotional barriers; tactics used by coercive men; practice. Unit 3 (Act) includes: assessing whether or not an escape is possible; research evidence on the effectiveness of resistance strategies; physical self-defense training. Unit 4 applies content to longer term relationships covering: comfort talking about sexuality, identification of sexual values, practices beyond intercourse, and articulation of relationship goals.
  Other Names: rape education
  Arms: Enhanced AAA Sexual Assault Education
Behavioral: Brochure — Current 'standard of care' at Canadian universities. Invitation to take and read brochures on sexual assault selected from those available on their Canadian university campus. All sites' brochures include general information on sexual assault and 'date-rape' drugs and post-rape legal and medical advice. The research assistant (RA) will ask the participants to take brochures, read them over, and to ask any questions they may have. Questions will be answered in a group setting and the participant will take home any brochures that she selected. Interaction between participants and the RA on the topic will be limited to 10-15 minutes and will be audio recorded for verification.
  Other Names: pamphlet
  Arms: Brochure

SUMMARY:
More than one in six women will be sexually assaulted in their lifetimes, most by men they know. The risk of sexual assault by men is greatest for girls and women between the ages of 14 and 24 making this a critical time for intervention. Sexual assault has many immediate and long-term negative consequences for victims. Even a small increase in the ability of women to resist sexual assault will result in a substantial improvement in the mental and physical health of women. Recent research has suggested that many young women delay their resistance to unwanted sexual advances because they are not sure that they are reading the situation correctly, they do not want to hurt the man's feelings, or they are unsure whether they have the right to say no to some sexual activity and say yes to other activity. Earlier work from the researchers resulted in the development of a program affecting these critical areas. This program was shown to be effective in helping participants build skills and a knowledge base to help them resist sexual assault and to prepare them for better recovery following sexual assault. The randomized controlled trial (RCT) builds on this prior work. We will establish whether the demonstrated short term effectiveness of this theoretically and empirically sound rape resistance intervention for university women extends to longer periods. We will determine whether the program can reduce the one year incidence of sexual assault by 30% among women attending Canadian universities. The results will also be used to indicate how long the effects of the program last and will indicate at which point in time refresher sessions may be necessary. A lay summary of the findings of the trial with a focus on application will be provided to all Canadian universities and to Provincial/Territorial Ministries of Education. This will be followed up with contact with those most likely to be involved in current campus education efforts.

DETAILED DESCRIPTION:
Violence against women costs Canadians at least $1.5 billion each year in health related expenses (Day, 1995). The associated physical and mental health effects are extensive and the social and economic costs are staggering. The aim of this project is to reduce a very common form of violence against women, sexual assault, at Canadian universities. At least 1 in 6 women will experience an attempted or completed rape in their lifetimes (Tjaden & Thoennes, 2000). The situation on university campuses is even more startling with as many as 1 in 4 women experiencing rape or attempted rape while enrolled in university (Fisher, Cullen, & Turner, 2000). Reductions in sexual assault will have a direct impact on the mental and physical health of university women.

The proposed trial builds on the Principal Investigator's CIHR-funded research which developed, revised, and then tested the basic sexual assault resistance program against a non-random control. It also builds on the Ontario Women's Health Council funded RCT which evaluated the basic program against an enhanced version, and a no-program control. Our pilot work (N=214) revealed that women who had the program experienced lower rates of completed sexual assault (40 - 50% lower) at 3 and 6 months than women who did not. The program also produced measurable improvements in knowledge, attitudes, and skills related to sexual assault resistance and to better recovery following sexual assault. This testing was within one university setting and with only short-term (1 week,3 and 6 month post) follow-up. This RCT extends this evaluation by expanding the participant population and examining the longer term efficacy of the program. First year female students from three Canadian universities will be randomized to receive our education program or to be part of a current practice exposure condition. Outcome measures will be completed at baseline, 1 week, 6, 12 months.

The four session sexual assault resistance program under study is based on the best theories and evidence available.Three of the four sessions address steps in a woman's emotional and cognitive processes as they relate to male acquaintances who are acting in a way that makes sexual coercion or sexual assault more likely. The units provide information, skills, and practice aimed at a) decreasing the time needed for women to assess the situation as dangerous and take action, b) reducing emotional obstacles to taking action, and c) increasing the use of the most effective methods of verbal and physical self-defense. The enhanced program piloted in the OWHC project includes a fourth unit which focuses on facilitating a stronger positive sexuality from which women may resist sexual coercion by male intimates more successfully.

The primary objective of this study is to establish whether a novel, small-group education program can reduce the one-year incidence of sexual assault by 30% (absolute difference of 7.5%). The secondary objectives are to assess whether changes in knowledge, attitudes, and skills related to the process of sexual assault resistance are improved in the short term, and, along with the primary outcome, maintained for the longer term. The tertiary objective is to assess whether the education program can also reduce the one-year incidence of forced sexual contact and sexual coercion.

The results of the trial will be used either to: (a) produce a maximally effective rape resistance education program package which can be adopted by universities across Canada or; (b) provide direction for further research into which aspects of the program need to be strengthened before such broad dissemination. The results will also be used to indicate how long the effects of the program last and will indicate at which point in time refresher sessions may be necessary.

ELIGIBILITY:
Inclusion Criteria:

* female subjects, aged 18 to 24 years;
* first-year university student;
* provide informed consent;
* able to attend one of four scheduled programs in the semester they are enrolled.

Exclusion Criteria:

None

Ages: 17 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 916 (Actual)
Dates: Start 2011-09; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Time-to-event occurrence of completed sexual assault in one year since randomization | 12 months
  Completed sexual assault (rape) will have occurred when a participant indicates she has had at least one experience of threatened, forced, or drugged completed (not attempted) sexual activity (oral, anal, or vaginal intercourse - answered 'once' or more to any of 9 questions (2c, 2d, 2e, 3c, 3d, 3e, 4c, 4d, or 4e) in the period between the baseline measurement and the current day (Sexual Experiences Survey Short Form Victimization (SES-SFV)(Koss et al., 2007)

SECONDARY OUTCOMES:
Change from baseline in perception of risk of sexual assault by male acquaintances and maintenance to 6 and 12 months | baseline, 1 week post-intervention, 6 and 12 months
  Measured by one item ("What are your chances of being raped by someone you know?") adapted from Gray et al., (1990) and piloted extensively by Senn.
Change from baseline in women's perception of their ability to defend themselves if a sexual assault situation were to arise and maintenance at 6 and 12 months | baseline, 1 week and 6 and 12 months post-intervention
  Self-defense self-efficacy: Ozer & Bandura, 1990
Knowledge of effective rape resistance strategies | 1 week post-intervention
  number of forceful physical and forceful verbal strategies in response to threatening hypothetical situations (Resistance measure, Testa et al., 2006; qualitative items by Senn) and real situations (items requesting details following sexual assaults experienced, questions added to SES items, Hanson & Gidycz, 1993).
Ability to realistically assess risk of harm in hypothetical scenarios where acquaintance sexual assault is likely | 1 week post-intervention
  A) Risk perception questionnaire (Testa et al., 2006). B) Risk Perception Survey (RPS) (Messman-Moore & Brown, 2006)
Change from baseline in beliefs and attitudes about rape | baseline, 1 week, 6 and 12 months post-intervention
  Indicated by endorsement of rape myths (Illinois Rape Myth Acceptance Scale (IRMA-SF), Payne, et al., 1999) and misinformation about the causes of rape (Perceived Causes of Rape Scale (PCOR), Cowan & Campbell, 1995; revised Cowan & Quinton, 1997); focus on Female Precipitation subscale.
Time-to-event occurrence of forced sexual contact and/or sexual coercion in one year since randomization | 12 months
  Using the SES-SFV, forced sexual contact will have occurred when a participant indicates she has had an experience of threatened, forced, or drug facilitated sexual touch not including intercourse - answered 'once' or more to any of 3 questions (1c, 1d, or 1e). Sexual coercion will have occurred when a participant reports one or more incidents of verbally coerced (excluding threats of physical harm) non-consensual oral, vaginal, or anal intercourse - answered 'once' or more to any of 6 questions (2a, 2b, 3a, 3b, 4a, or 4b) in the period between the baseline measurement and the current day.
Maintenance of improved knowledge of effective rape resistance strategies | 12 months
  number of forceful physical and forceful verbal strategies in response to threatening hypothetical situations (Resistance measure, Testa et al., 2006; qualitative items by Senn) and real situations (items requesting details following sexual assaults experienced, questions added to SES items, Hanson & Gidycz, 1993).
Maintenance of ability to realistically assess risk of harm in hypothetical scenarios where acquaintance sexual assault is likely | 12 months
  A) Risk perception questionnaire (Testa et al., 2006). B) Risk Perception Survey (RPS) (Messman-Moore & Brown, 2006)

CONTACTS AND LOCATIONS:
Overall Officials: Charlene Y Senn, PhD, Principal Investigator — University of Windsor
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Guelph, Guelph, Ontario

REFERENCES:
- [Background] Senn CY, Gee S & Thake J. Emancipatory sexuality education and sexual assault resistance: Does the former enhance the latter? Psychology of Women Quarterly 35(1): 72-91, 2011.
- [Background] Day, T. (1995). The Health-Related Costs of Violence against Women in Canada: The Tip of the Iceberg. London, On.: The Centre for Research on Violence Against Women and Children, 1995.
- [Background] Tjaden P, Thoennes N. Full Report of the Prevalence, Incidence, and Consequences of Violence Against Women: Findings From the National Violence Against Women Survey. U.S. Department of Justice Office of Justice Programs, 2000.
- [Background] Fisher B, Cullen F, Turner M. The Sexual Victimization of College Women: Findings From Two National-Level Studies. Washington, DC: National Institute of Justice and Bureau of Justice Statistics, 2000.
- [Background] Koss MP, Abbey A, Campbell R, Cook S, Norris J, Testa M. et al. Revising the SES: A collaborative process to improve assessment of sexual aggression and victimization. Psychology of Women Quarterly, 31(4), 357-370, 2007.
- [Background] Ozer EM, Bandura A. Mechanisms governing empowerment effects: a self-efficacy analysis. J Pers Soc Psychol. 1990 Mar;58(3):472-86. doi: 10.1037//0022-3514.58.3.472. PMID 2324938
- [Background] Gray DM, Lesser D, Quinn E, Brounds C. The effectiveness of personalizing acquaintance rape prevention: Programs on perception of vulnerability and on reducing risk-taking behavior. Journal of College Student Development, 31, 217-220, 1990.
- [Background] Hanson KA, Gidycz CA. Evaluation of a sexual assault prevention program. J Consult Clin Psychol. 1993 Dec;61(6):1046-52. doi: 10.1037//0022-006x.61.6.1046. PMID 8113482
- [Background] Testa M, Vanzile-Tamsen C, Livingston JA, Buddie AM. The role of women's alcohol consumption in managing sexual intimacy and sexual safety motives. J Stud Alcohol. 2006 Sep;67(5):665-74. doi: 10.15288/jsa.2006.67.665. PMID 16847534
- [Background] Messman-Moore TL, Brown AL. Risk perception, rape and sexual revictimization: A prospective study of college women. Psychology of Women Quarterly, 30, 159-172, 2006.
- [Background] Payne DL, Lonsway KA, Fitzgerald LF. Rape myth acceptance: Exploration of its structure and its measurement using the Illinois Rape Myth Acceptance Scale. Journal of Research in Personality, 33, 27-68, 1999.
- [Background] Cowan G, Campbell RR. Rape causal attitudes among adolescents. Journal of Sex Research, 32, 145-153, 1995.
- [Background] Cowan G, Quinton WJ. Cognitive style and attitudinal correlates of the perceived causes of rape scale. Psychology of Women Quarterly, 21, 227-245, 1997.
- [Derived] Hobden KL, Thurston WE, McVey GL, Senn CY. An Evaluation of Strategies Used to Maximize Intervention Fidelity in a Randomized Controlled Trial of a Sexual Assault Resistance Program for University Women. Prev Sci. 2021 Oct;22(7):960-970. doi: 10.1007/s11121-021-01239-2. Epub 2021 Apr 17. PMID 33864584
- [Derived] Senn CY, Eliasziw M, Barata PC, Thurston WE, Newby-Clark IR, Radtke HL, Hobden KL. Efficacy of a sexual assault resistance program for university women. N Engl J Med. 2015 Jun 11;372(24):2326-35. doi: 10.1056/NEJMsa1411131. PMID 26061837
- [Derived] Senn CY, Eliasziw M, Barata PC, Thurston WE, Newby-Clark IR, Radtke HL, Hobden KL; SARE Study Team. Sexual violence in the lives of first-year university women in Canada: no improvements in the 21st century. BMC Womens Health. 2014 Nov 5;14:135. doi: 10.1186/s12905-014-0135-4. PMID 25410412
- [Derived] Senn CY, Eliasziw M, Barata PC, Thurston WE, Newby-Clark IR, Radtke HL, Hobden KL; SARE study team. Sexual assault resistance education for university women: study protocol for a randomized controlled trial (SARE trial). BMC Womens Health. 2013 May 23;13:25. doi: 10.1186/1472-6874-13-25. PMID 23702221